CLINICAL TRIAL: NCT07098390
Title: The Effect of Progressive Muscle Relaxation Exercise Undergoing Total Hip and Knee Arthroplasty Patients on Fear of Falling, Pain and Anxiety Level
Brief Title: Effect of Progressive Muscle Relaxation on Fear of Falling, Pain, and Anxiety in Arthroplasty Patients
Acronym: PMRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Zühal Erdoğan, Gazi University, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025 - 1072
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Arthoplasty, Pain, Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Since the progressive muscle relaxation exercise (PMRE) is administered by the researcher in this study, blinding of the researcher will not be possible. However, to ensure participant blinding, PMRE will be provided to the control group after the final assessments are completed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation Exercise (Experimental)
  Interventions: Behavioral: Progressive Muscle Relaxation Exercise
- Control (No Intervention): Participants in this group will receive routine perioperative care

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation Exercise — When patients are admitted to the Orthopedics and Traumatology Clinic for arthroplasty and agree to participate in the study, they will be informed about the research process and written informed consent will be obtained. The Descriptive Information Form, Numeric Rating Scale (NRS), The Fear of Falling Scale, and the State-Trait Anxiety Inventory (STAI) will be administered through face-to-face interviews by the researcher. After the pre-tests are completed, patients will be randomly assigned to the intervention and control groups.
  In the preoperative period, upon admission to the clinic, patients in the intervention group will receive progressive muscle relaxation exercises (PMRE). To enhance concentration and minimize the impact of ambient noise, patients will listen to the exercises using headphones.
  On the first postoperative day, the patient will be revisited by the researcher. After the physician explains that the patient will be mobilized, the State-Trait Anxiety Inventory will
  Arms: Progressive Muscle Relaxation Exercise

SUMMARY:
The study will be conducted using a parallel-group randomized controlled experimental design to determine the effect of progressive muscle relaxation exercises on postoperative fear of falling, pain, and anxiety levels in patients undergoing total hip and knee arthroplasty. The study group will consist of patients who have undergone total hip or knee arthroplasty in the Orthopedics and Traumatology Clinic of a university hospital.

Research data will be collected using the "Descriptive Information Form," the The Fear of Falling Scale, the Numeric Rating Scale (NRS), and the State-Trait Anxiety Inventory. Patients will be randomly assigned to intervention and control groups, and progressive muscle relaxation exercises will be applied to the patients in the intervention group.

DETAILED DESCRIPTION:
When patients are admitted to the Orthopedics and Traumatology Clinic for arthroplasty and agree to participate in the study, they will be informed about the research process and written informed consent will be obtained. The Descriptive Information Form, Numeric Rating Scale (NRS), The Fear of Falling Scale, and the State-Trait Anxiety Inventory (STAI) will be administered through face-to-face interviews by the researcher. After the pre-tests are completed, patients will be randomly assigned to the intervention and control groups.

In the preoperative period, upon admission to the clinic, patients in the intervention group will receive progressive muscle relaxation exercises (PMRE). To enhance concentration and minimize the impact of ambient noise, patients will listen to the exercises using headphones.

On the first postoperative day, the patient will be revisited by the researcher. After the physician explains that the patient will be mobilized, the State-Trait Anxiety Inventory will be administered, and the patient's pain and fear of falling will be evaluated. PMRE will then be performed, followed by the patient's first mobilization. One hour after mobilization, fear of falling, state-trait anxiety, and pain will be reassessed. The PMRE sessions, lasting approximately 30 minutes, will be guided with slow and rhythmic instructions, delivered in a soft tone of voice and accompanied by music.

For patients in the control group, the administration of the questionnaires will be conducted in the same manner as in the intervention group. Upon admission to the clinic, the Descriptive Information Form, Numeric Rating Scale (NRS), The Fear of Falling Scale, and the State-Trait Anxiety Inventory will be completed through face-to-face interviews. On the first postoperative day, the patient will be revisited by the researcher, and after the physician explains that the patient will be mobilized, the State-Trait Anxiety Inventory will be administered again, and the patient's pain and fear of falling will be evaluated. The patient's first mobilization will then be carried out. One hour after mobilization, fear of falling, state-trait anxiety, and pain will be reassessed.

Pain assessment will begin from the second postoperative hour. Pain intensity will be evaluated every 2 hours for the first 8 hours and then every 4 hours thereafter. After the final assessments of the control group are completed, PMRE will be administered by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18 years or older,

  * Undergoing primary and elective hip or knee arthroplasty,
  * Admitted to the clinic one day before surgery,
  * Having no other acute illness that could cause pain or anxiety,
  * Voluntarily agreeing to participate in the study,
  * Able to communicate

Exclusion Criteria:

* • Diagnosed with any neurological or psychiatric disorder affecting cognitive status,

  * Diagnosed with an anxiety disorder,
  * Developing complications during the perioperative period,
  * Undergoing active cancer treatment,
  * Receiving chronic pain treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
The Fear of Falling Scale | Baseline Twice a day on the first postoperative day
  The Fear of Falling Scale consists of a single-item question asking participants to indicate their fear of falling on a four-point Likert scale: 1 = not afraid, 2 = slightly afraid, 3 = moderately afraid, and 4 = very afraid. This scale has been widely used in various studies, particularly among patients with hip fractures (Damar et al., 2018).
Numeric Rating Scale (NRS): | Baseline Pain assessment will begin at the 2nd hour after surgery. During the first 8 hours, pain intensity will be evaluated every 2 hours, and then every 4 hours thereafter.
  The Numeric Rating Scale is a unidimensional tool designed to assess the intensity of pain, allowing patients to express their pain using numbers. It is an 11-point scale ranging from 0 (no pain) to 10 (unbearable pain). Scores of 1-3 indicate mild pain, 4-6 indicate moderate pain, and 7-10 indicate severe pain. It is a valid and reliable tool for assessing postoperative pain in conscious patients
State-Trait Anxiety Inventory (STAI): | Baseline Twice a day on the first postoperative day
  The State-Trait Anxiety Inventory (STAI), developed by Spielberger et al. to measure individuals' levels of state and trait anxiety, was adapted into Turkish and validated by Öner and Le Compte (1977). The scale evaluates how individuals feel about themselves and consists of two subscales, both using a four-point Likert format.
  The first part, the State Anxiety Scale, includes 20 items and assesses how the individual feels at a specific moment and under specific conditions (Öner, 1985).
  The second part, the Trait Anxiety Scale, also includes 20 items and measures the individual's general tendency to experience anxiety. It was developed to reflect the anxiety experienced over the past seven days. Some items are reverse-scored when calculating the total score. In the State Anxiety Scale, 10 items (1, 2, 5, 8, 10, 11, 15, 16, 19, 20) are reversed; in the Trait Anxiety Scale, 7 items (21, 26, 27, 30, 33, 36, 39) are reversed.
  After reversing the scores of negatively worded items, the tota

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)